CLINICAL TRIAL: NCT02013089
Title: A Pilot Study of Genomic Sequencing Guided Individualized Therapy in Gastrointestinal Cancers
Brief Title: A Pilot Study of Genomic Sequencing Guided Individualized Therapy in Gastrointestinal Cancers, GITIC Study
Acronym: GITIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Associate Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU04
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Gastrointestinal Cancers
Keywords: genomic sequencing, Integrated genomic network analysis
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Erlotinib Hydrochloride; Gefitinib; Everolimus; Imatinib Mesylate; Sorafenib; Sunitinib; vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Erlotinib or Gefitinib (Experimental): Erlotinib 150 mg tablet or Gefitinib 250 mg tablet by mouth every day
  Interventions: Drug: Erlotinib or Gefitinib
- Everolimus (Experimental): Everolimus 10 mg orally once daily every day
  Interventions: Drug: Everolimus
- Imatinib (Experimental): Imatinib 400 mg tablet orally per day
  Interventions: Drug: Imatinib
- Sorafenib or Sunitinib (Experimental): Sorafenib 400 mg twice a day at least one hour before or two hours after eating or Sunitinib 50 mg orally once a day
  Interventions: Drug: Sorafenib or Sunitinib
- Vandetanib (Experimental): Vandetanib 300 mg orally once daily
  Interventions: Drug: Vandetanib
- Control (No Intervention): No intervention was performed for patients without any gene alternation or without any available target agents

INTERVENTIONS:
Drug: Erlotinib or Gefitinib — Erlotinib 150mg talbet or Gefitinib 250 mg tablet per day for patients with EGFR gene alternation
  Other Names: Erlotinib (Tarceva®) or Gefitinib (Iressa®)
  Arms: Erlotinib or Gefitinib
Drug: Everolimus — Everolimus 10 mg orally once daily every day for patients with mTOR gene alternation
  Other Names: Afinitor®
  Arms: Everolimus
Drug: Imatinib — Imatinib 400 mg tablet orally per day for patietns with KIT, PDGFR, ABL gene alternation
  Other Names: Gleevec®
  Arms: Imatinib
Drug: Sorafenib or Sunitinib — Sorafenib 400 mg twice a day at least one hour before or two hours after eating or Sunitinib 50 mg orally once a day with or without food for patients with VEGFR, KIT, RAF gene alternation
  Other Names: Sorafenib (Nexavar®) Sunitinib (Sutent®)
  Arms: Sorafenib or Sunitinib
Drug: Vandetanib — Vandetanib 300 mg orally once daily for patients with RET gene fusion.
  Other Names: Caprelsa®
  Arms: Vandetanib

SUMMARY:
Hypothesis: Different patients have different biomarkers, if doctors know about the biomarkers of patients; they may be able to prescribe a regimen that is better suited to the patient's specific needs. This is a pilot study. Here, we used whole exon sequencing and Integrated genomic network analysis to identify the biomarker or gene. We aimed to learn if the drug chosen based on biomarkers can help to control metastatic gastrointestinal cancer who had failed from all standard and available regimens.

DETAILED DESCRIPTION:
Rational: Cancer sequencing (CS) promises to become the centerpiece of personalized oncology by informing on treatments targeted to each tumor's unique genetic constitution. This data can be critical to making an informed decision for disease management, though this may not be the case for all patients. CS identifies variations or differences in the DNA and/or RNA of the cells in an individual's tumor by comparison to that of his/her normal cells. These somatic variations may, on further interpretation, be identified as key drivers of carcinogenesis. Such information may predict a patient's prognosis, response to currently available treatments or prompt the development of novel therapeutics. Though CS has the potential to personalize and optimize cancer care, it may produce a vast amount of data and unique changes in the DNA/RNA that may be difficult to interpret at the present time.

Using the Integrated genomic network analysis, we could have better understanding of the underlying processes and pathways involved in tumor onset and progression. And then we could choose a specific treatment regimen and develop personalized cancer therapies

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic diagnosis of Gastrointestinal cancer
2. The subject has a diagnosis metastatic gastrointestinal cancer, and failed from standard treatment, and no other regimen is available.
3. The subject has measurable lesion of gastrointestinal cancer.
4. The subject's The Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. The subject has adequate hematologic function as defined by an absolute neutrophil count (ANC) >/= 1,500/mm3, platelet count >/= 100,000/mm3, White Blood Count (WBC) >/= 3,000/ mm3, and hemoglobin >/= 9 g/dL.
6. The subject has adequate hepatic function as defined by a total bilirubin level </= 1.5 * the upper limit of normal (ULN) (bilirubin >/= 1.5 * ULN with known Gilbert's disease is allowed), and alkaline phosphatase, aspartate aminotransferase/alanine aminotransferase (AST/ALT) </= 2.5 * the upper limit of normal or </= 5.0 * ULN if liver metastases are present.
7. Serum creatinine clearance >50ml/min, either by Cockcroft-Gault formula or 24-hour urine collection analysis
8. The subject is >/=18 years of age.
9. The subject has signed informed consent.
10. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Childbearing potential will be defined as women who have had menses within the past 12 months, who have not had tubal ligation, hysterectomy or bilateral oophorectomy. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

1. pregnant or breast-feeding.
2. Subjects will be excluded for other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study
3. without enough tumor sample for analysis.
4. Refuse to sign the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  From the date of enrollment until the date of death from any cause.

SECONDARY OUTCOMES:
Response rate | 1 year
  After identifying the driver gene and choosing the specific target drug, the response rate of all patients.

OTHER OUTCOMES:
Disease control rate | 1 year
  The disease control rate of all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yanghong Deng, PhD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China